CLINICAL TRIAL: NCT06026423
Title: Dehisced Perineal Tear After Vaginal Labour (HEAL) - Conservative Treatment or Resuturing
Brief Title: Conservative Treatment or Resuturing Among Women With Perineal Wound Dehiscence After Vaginal Labour
Acronym: HEAL
Status: Recruiting | Type: Observational
Sponsor: Herlev Hospital (Other)
Responsible Party: Principal Investigator, Hanna Jangö, Staff specialist, Ph.D., Associated professor, Herlev Hospital
Other Study IDs: H-23022460
Record Dates: First submitted 2023-08-30; First posted 2023-09-07 (Actual); Last update posted 2023-09-18 (Actual); Status verified 2023-09

CONDITIONS: Dehiscence Wound; Secondary Perineal Tear; Episiotomy; Dehiscence
Keywords: Dehiscence; Secondary Perineal Tear; Episiotomy
MeSH Terms: interventions — Restraint, Physical; Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Normal/uncomplicated healing process: 100 women with a second-degree tear or episiotomy primarily sutured after labor: identified with a normal/uncomplicated healing process
  Interventions: Other: Clinical examination and pictures; Other: Questionnaire
- Dehisced wound treated with secondary resuturing: 100 women with a second-degree tear or episiotomy: identified with a dehisced wound treated with secondary resuturing
  Interventions: Other: Clinical examination and pictures; Other: Questionnaire
- Dehisced wound treated with conservative management: 100 women with a second-degree tear or episiotomy: identified with a dehisced wound treated with conservative management
  Interventions: Other: Clinical examination and pictures; Other: Questionnaire

INTERVENTIONS:
Other: Clinical examination and pictures — A clinical examination is needed to assess the healing process for the three groups. After assessing the healing process, we will take pictures of the tear for documentation.
Other: Questionnaire — The participant will answer questions, serving as a baseline questionnaire, when arriving at the clinical examination one month post-partum. At three and 9-12 months post-postpartum, they will receive another questionnaire. The questionnaire will consist of validated questions regarding body image, pain, Urogynecological problems as symptoms of prolapse, urinary and anal incontinence, and questions about sexual problems.

SUMMARY:
The goal of this observational study is to make us more aware of the short and long-term outcomes for women having an uncomplicated healing process after a rupture or birth cut in the perineum after giving birth in relation to a healing process with a dehisced wound treated with conservative management or secondary suturing.

Participants will be asked to do

* A gynecological examination at one month after birth and 9-12 months after birth.
* Have a picture taken of the healing process
* Answer a questionnaire at one month, three months, and 9-12 months after birth

DETAILED DESCRIPTION:
The best way to manage perineal wound dehiscence after childbirth is unknown. Currently, there is no agreed best practice recommendation for managing perineal wound dehiscence due to a lack of evidence comparing conservative management with secondary suturing. Therefore, studies are urgently needed to compare the benefits and risks of both treatments. This study has the potential to significantly impact women´s health for those suffering from perineal wound dehiscence.

The investigators want to include 100 women who have had a primary repair of a second-degree tear or episiotomy with a normal/uncomplicated healing process, 100 women with a second-degree tear or episiotomy identified with a dehisced wound treated with secondary resuturing, and 100 women with a second-degree tear or episiotomy identified with a dehisced wound treated with conservative management.

All women who meet the inclusion criteria are recommended the same treatment and follow-up as currently present as standard care at the four hospitals that the investigators are recruiting from. The study deviates from the standard of care by offering two extra clinical examinations, one questionnaire evaluation without clinical examination, and a follow-up with pictures of the perineal tear healing process.

ELIGIBILITY:
Inclusion Criteria:

* Women with a vaginal delivery who have had a primary repair of a second-degree perineal tear or episiotomy
* At least 18 years old
* Able to understand, read and speak Danish or English
* Able to give informed consent

Exclusion Criteria:

* None, first, third- and fourth-degree tear
* Cesarean Section

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: We want to include 100 women who have had a primary repair of a second-degree tear or episiotomy with an uncomplicated healing process. They will only be recruited from the Perineal Care Clinics at the Department of Obstetrics and Gynecology at the Copenhagen University Hospital - Herlev. Furthermore, we want to include 100 women with a second-degree tear or episiotomy identified with a dehisced wound treated with secondary resuturing, and 100 women with a second-degree tear or episiotomy identified with a dehisced wound treated with conservative management. They will be recruited from the Perineal Care Clinics at the Department of Obstetrics and Gynecology at the Copenhagen University Hospitals - Rigshospitalet, Herlev Hospital, North Zealand Hospital, and Hvidovre Hospital. The women will come for a clinical examination to assess wound infection and healing 4 - 14 days post-partum.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-09-15 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Body image | 9-12 months
  Measured by the Body-Image questionnaire FGSIS - Female Genital Self-Image Scale

SECONDARY OUTCOMES:
Wound healing | One month
  The proportion of women with healed wounds at one month post-partum assessed by clinical examination and REEDA scale (Redness, Oedema, Ecchymosis, Discharge, Approximation of the wound edges). The REEDA scale contains five criteria each receiving a score between 0 and 3. The total score range from 0 - 15 with lower scores representing better-wound healing
Infection rate | One month
  The proportion of women with an infected wound until one month post-partum assessed by clinical examination and measured by REEDA scale
Resuming sexual intercourse | One month, three months, and 9-12 months
  Measured by the PISQ-12 questionnaire which is a short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12)
Dyspareunia | One month, three months, and 9-12months
  Measured by the PISQ-12 questionnaire which is a short form of the Pelvic Organ Prolapse/Urinary Incontinence Sexual Questionnaire (PISQ-12)
Woman´s satisfaction with the aesthetic results of the perineal wound | One month, three months, and 9-12 months
  Self-reported. The woman will be asked if she is satisfied with the aesthetic results of the perineal wound
Affected breastfeeding | One month, three months, and 9-12 months
  The woman will be asked whether she is breastfeeding or not
Re-admission | Within one month
  The women will be asked whether they have been readmitted to the hospital and why within four weeks p.p.
Prolapse | One month, three months, and 9-12 months
  Measured by ICIQ-VS questionnaire which is a short form of the International Consultation on Incontinence Questionnaire - Vaginal Symptoms (ICIQ-VS)
Urinary incontinence | One month, three months, and 9-12 months
  Measured by the ICIQ-UI SF questionnaire which is a short form of the International Consultation on Incontinence Questionnaire - Urinary Incontinence Short Form (ICIQ-UI SF)
Fecal incontinence | One month, three months, and 9-12 months
  Measured by ICIQ-B questionnaire which is a short form of the International Consultation on Incontinence Questionnaire - Bowel (ICIQ-B)
Psychological well-being (maternal anxiety or depression) | Three months, and 9-12 months
  Measured by Edinburgh Postnatal Depression Scale (EPDS). EPDS is a self-assessment questionnaire consisting of ten statements and the respondent is asked about their feelings over the last seven days. The answers are scored from 0-3 which gives an endpoint from 0-30. In Denmark, women are said to have depressive symptoms after delivery if they score 11 or higher
Pain intensity | One month, three months, and 9-12 months
  Self-reported pain intensity measured by Visual Analog Scale (VAS-score). Numeric rating scale from 0-10 (0 = no pain - 10 = pain as bad as can be)
Consuming painkillers because of pain due to perineal tear | One month, three months, and 9-12 months
  The participant will be asked whether she is consuming painkillers because of pain due to a perineal tear (Yes/No)
Pelvic floor muscle contraction | One month and 9-12 months
  Measured by Modified Oxford scale

CONTACTS AND LOCATIONS:
Overall Officials: Hanna M. Jangö, MD, PhD, Principal Investigator — Copenhagen University Hospital - Herlev and Gentofte
Locations (1):
- Department of Obstetrics and Gynaecology, Copenhagen University Hospital - Herlev and Gentofte, Herlev, Denmark

IPD SHARING:
Plan to Share IPD: Undecided